CLINICAL TRIAL: NCT04468841
Title: An Exploratory Study to Correlate the Level of Cell-free DNA With Response to First-line Treatment in Patients With Follicular Lymphoma
Brief Title: Measuring Cell-Free DNA (cfDNA) Levels in People With Follicular Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-199
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Follicular Lymphoma
Keywords: Cell-free DNA; 20-199
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: This is a non-therapeutic protocol. The intervention in this study will involve collection of a standard-of-care pre-treatment tumor biopsy (archival tissue, if available) to identify the tumor-specific s cfDNA signature.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Group (Experimental): Study participants with untreated, newly diagnosed follicular lymphoma will have blood collected for cfDNA testing before, during, and after their first-line treatment or observation period
  Interventions: Diagnostic Test: cfDNA testing; Other: sample of saliva or fingernail clipping; Diagnostic Test: pre-treatment test specimen; Diagnostic Test: PET/CT, CT, or MRI testing
- Retrospective Group (Experimental): Study participants who have received first-line treatment for follicular lymphoma and are in complete remission will have blood collected for cfDNA testing. In the retrospective cohort, MSKCC patients with CRs lasting ≥10 years after induction therapy will be studied. Initial tumor tissue (if available) will be collected to examine the status of s cfDNA in patients with long-term remissions. Blood samples will be collected once, if the patient has interesting results (e.g. positive cfDNA sample despite CR on imaging, etc.) then additional blood samples may be taken during follow up visits.
  Interventions: Diagnostic Test: cfDNA testing; Other: sample of saliva or fingernail clipping; Diagnostic Test: pre-treatment test specimen; Diagnostic Test: PET/CT, CT, or MRI testing

INTERVENTIONS:
Diagnostic Test: cfDNA testing — peripheral blood samples collected before initiation of standard therapy, after 2 cycles of therapy, at the completion of 6-8 cycles of induction therapy, and then every 6 months for a total of 2 years from the initiation of therapy using a cfDNA assay. For retrospective patients, blood samples will be collected once.
Other: sample of saliva or fingernail clipping — collected in clinic one time
Diagnostic Test: pre-treatment test specimen — From bone marrow, blood, lymph node, or alternate site to identify tumor-specific mutations. For retrospective patients initial tumor tissue (if available).
Diagnostic Test: PET/CT, CT, or MRI testing — PET/CT scans are required at baseline and at the patient's end-of-treatment visit. The other standard-of-care scan timepoints can be performed using PET/CT, dedicated CT, or MRI per the treating investigator's discretion.

SUMMARY:
The researchers are doing this study to measure and test cell-free DNA (cfDNA) in the blood before, during, and after first-line treatment for follicular lymphoma. They will look at whether cfDNA levels are related to a person's response to the usual first-line treatment for follicular lymphoma. Researchers also want to understand how different genetic changes in follicular lymphoma relate to a person's response to the usual first-line treatment.

DETAILED DESCRIPTION:
This is a non-therapeutic protocol aimed to assess the ability of the s cfDNA assay to detect clinical response in FL when compared to conventional approaches for assessing response, such as PET-CT scans.

Study assessments will include: 1) identification of the mutations present in the primary tumor, 2) identification of these mutations in the peripheral blood samples collected before initiation of standard therapy, after 2 cycles of therapy, at the completion of 6-8 cycles of induction therapy, and then every 6 months for a total of 2 years from the initiation of therapy using a cfDNA assay. For patients who receive RT, peripheral blood samples will be collected before initiation of RT, and then 3 months, 6 months, 12 months, 18 months and 24 months post RT using a s cfDNA assay.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at time of signing informed consent. Consent is permitted from either the participant or from a Legally Authorized Representative (LAR) on their behalf.
* Histology-confirmed follicular lymphoma grade 1-3a, verified by the enrolling institution
* Ability to adhere to the study visit schedule and all the protocol requirements
* Measurable FDG-avid disease
* Not applicable for retrospective patients in CR

Exclusion Criteria:

* Patients receiving second or greater line of therapy (except in retrospective cohort of long-term survivors of FL [i.e. >10 years out from frontline treatment])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
whether the assay can correctly identify presence of disease in patients with measurable disease | 2 years
  Response will be evaluated using the updated response criteria entitled, "The Lugano Classification" system. The investigator will use of the 5-point scale for visually assessing response on the pre- and end-of-treatment FDGPET/CT scans. This scale is commonly referred to as the Deauville criteria; it was developed by international experts in the field at the First International Workshop on interim-PET in Lymphoma in Deauville in 2009 and is routinely applied to patients undergoing lymphoma directed therapy. The 5-point scale is described in the table below.
  1 No residual uptake 2 Uptake ≤ mediastinum 3 Uptake > mediastinum but ≤ liver 4 Uptake moderately > liver 5 Markedly increased uptake at any site or progression

CONTACTS AND LOCATIONS:
Overall Officials: Paola Ghione, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm